CLINICAL TRIAL: NCT07393932
Title: MND Together: Improving Communication and Coordination of Motor Neuron Disease Care
Brief Title: MND Together: Phase 1
Status: Not yet recruiting | Type: Observational
Sponsor: University of Sheffield (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Liverpool John Moores University (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Cornwall Partnership NHS Foundation Trust (Network); Northern Lincolnshire and Goole Hospitals NHS Foundation Trust (Other); Dementias Platform UK (Unknown); NIHR HealthTech Research Centre (Unknown); Swansea Bay University Health Board (Other)
Responsible Party: Sponsor
Other Study IDs: R/186866
Record Dates: First submitted 2026-01-15; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: MND (Motor Neurone DIsease)
Keywords: MND; Care coordination; health and social care; multidisciplinary care; community services; Motor Neurone Disease; Neurological conditions; ethnography; Amyotrophic lateral sclerosis (ALS); Qualitative
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable- observational study — MND-Together tool will be informed by the findings from this study

SUMMARY:
This project consists of two workstreams, both of which will be mixed-methods and aim to develop a national UK picture of current care coordination for people with MND, including observations of barriers and facilitators. The studies will explore how care is transferred and communicated across MND specialist services to non-specialist community health settings.

In workstream 1, the researchers will conduct focus groups with people with MND, Carers, former Carers, Health and Social Care Professionals and managers and commissioners. These focus groups, alongside the analysis of routine data, will create a national picture of MND care and begin a behavioural diagnosis of the barriers and facilitators. In workstream 2, a multi-site ethnography study will be conducted, including observations, interviews, routine data, care plan and document review. This Workstream will observe how care is coordinated between specialist and non-specialist services and continue to explore barriers and facilitators that can not be identified through interviews.

ELIGIBILITY:
WS1

Inclusion Criteria:

* Person with MND, carers, former carers, Health and Social Care Professionals, managers and commissioners
* Ability to engage in focus group or interview or email interview

Exclusion Criteria:

* no exclusion criteria

WS2

Inclusion Criteria:

* Person with MND, carers, former carers, Health and Social Care Professionals, managers and commissioners
* Ability to engage in an observations and interviews

Exclusion Criteria:

* no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People attending MND specialist centres and non specialist community services
Sampling Method: Non-Probability Sample
Enrollment: 287 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of barriers and facilitators for capability, opportunity and motivation (COM-B) | February 2026- February 2027

CONTACTS AND LOCATIONS:
Overall Officials: Liam Knox, PhD, Principal Investigator — University of Sheffield; Chris McDermott, MBChB, FRCP, PhD, Principal Investigator — University of Sheffield
Locations (1):
- School of Medicine and Populational Health, Sheffield, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The pseudo-anonymised data, and analysis output will be uploaded to the University of Sheffield data repository, ORDA, and stored for 10 years as per the University of Sheffield Retention Schedule. The data will be embargoed until the study has been published in a peer-reviewed journal and will be available thereafter to other researchers upon reasonable request to the CI.
Time Frame: After the study has been published in a peer-review journal and it will be kept on the data repository for 10 years